CLINICAL TRIAL: NCT02974361
Title: An Open-label, Single-dose, Randomised, Crossover Study to Evaluate Changes in the Pharmacokinetics of Ibuprofen From Ibuprofen-LDH Dosed With and Without Release Modifying Excipients in Normal, Healthy, Adult Subjects
Brief Title: Impact of Excipients on Pharmacokinetics of OXPzero(TM) Ibuprofen
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oxford Pharmascience Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: OAT-01
Record Dates: First submitted 2016-11-21; First posted 2016-11-28 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Pharmacokinetics
MeSH Terms: interventions — Ibuprofen

ARMS (17):
- Part A Ibuprofen control (Active Comparator)
  Interventions: Drug: Ibuprofen
- Part A Ibuprofen-LDH (Experimental)
  Interventions: Drug: Ibuprofen-LDH
- Part A Ibuprofen-LDH Excipient Combo 1 (Experimental)
  Interventions: Drug: Ibuprofen-LDH
- Part A Ibuprofen-LDH Excipient Combo 2 (Experimental)
  Interventions: Drug: Ibuprofen-LDH
- Part A Ibuprofen-LDH Excipient Combo 3 (Experimental)
  Interventions: Drug: Ibuprofen-LDH
- Part A Ibuprofen-LDH Excipient Combo 4 (Experimental)
  Interventions: Drug: Ibuprofen-LDH
- Part A Ibuprofen Lysine (Active Comparator)
  Interventions: Drug: Ibuprofen Lysine
- Part B Ibuprofen (Active Comparator)
  Interventions: Drug: Ibuprofen
- Part B Ibuprofen LDH Excipient Combo 1 (Experimental)
  Interventions: Drug: Ibuprofen-LDH
- Part B Ibuprofen LDH Excipient Combo 2 (Experimental)
  Interventions: Drug: Ibuprofen-LDH
- Part B Ibuprofen LDH Excipient Combo 3 (Experimental)
  Interventions: Drug: Ibuprofen-LDH
- Part B Ibuprofen LDH Excipient Combo 4 (Experimental)
  Interventions: Drug: Ibuprofen-LDH
- Part C Ibuprofen (Active Comparator)
  Interventions: Drug: Ibuprofen
- Part C Ibuprofen LDH Excipient Combo 1 (Experimental)
  Interventions: Drug: Ibuprofen-LDH
- Part C Ibuprofen LDH Excipient Combo 2 (Experimental)
  Interventions: Drug: Ibuprofen-LDH
- Part C Ibuprofen LDH Excipient Combo 3 (Experimental)
  Interventions: Drug: Ibuprofen-LDH
- Part B Ibuprofen LDH Excipient Combo 5 (Experimental)
  Interventions: Drug: Ibuprofen-LDH

INTERVENTIONS:
Drug: Ibuprofen
  Arms: Part A Ibuprofen control; Part B Ibuprofen; Part C Ibuprofen
Drug: Ibuprofen Lysine
  Arms: Part A Ibuprofen Lysine
Drug: Ibuprofen-LDH
  Arms: Part A Ibuprofen-LDH; Part A Ibuprofen-LDH Excipient Combo 1; Part A Ibuprofen-LDH Excipient Combo 2; Part A Ibuprofen-LDH Excipient Combo 3; Part A Ibuprofen-LDH Excipient Combo 4; Part B Ibuprofen LDH Excipient Combo 1; Part B Ibuprofen LDH Excipient Combo 2; Part B Ibuprofen LDH Excipient Combo 3; Part B Ibuprofen LDH Excipient Combo 4; Part B Ibuprofen LDH Excipient Combo 5; Part C Ibuprofen LDH Excipient Combo 1; Part C Ibuprofen LDH Excipient Combo 2; Part C Ibuprofen LDH Excipient Combo 3

SUMMARY:
This study is to help development of a new version of Ibuprofen, called Ibuprofen-LDH. Ibuprofen-LDH will be used as a treatment for muscular pains, headache, fever etc. This new version of ibuprofen is expected to produce fewer stomach/intestine related side effects when compared to many existing marketed formulations of Ibuprofen.

This study is split into 3 parts. Part A is a 7 way crossover, Part B is a maximum of a 6 way crossover and Part C is a maximum of a 4 way crossover. The size of Parts B & Part C and allocated interventions will be confirmed after review of data from Parts A and/or B respectively.

A total of 30 subjects will take part in the study; 10 per study part.

The key objective is to assess the pharmacokinetics properties of Ibuprofen-LDH, with and without a selection of different excipients. The pharmacokinetic properties will include how quickly the drug is absorbed into the bloodstream and also the maximum concentration of drug that reaches the bloodstream.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects
* BMI 18 - 30 kg/m2
* Willing and able to provide written informed consent

Exclusion Criteria:

* Evidence or history of significant renal, hepatic, gastrointestinal, central nervous system, respiratory, cardiovascular, autoimmune or metabolic dysfunction
* Recent or concurrent use of prescription or non-prescription medications, other than contraceptives
* Allergy or sensitivity to NSAIDs

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-12; Primary Completion 2017-04-28 (Actual); Study Completion 2017-05-03 (Actual)

PRIMARY OUTCOMES:
Cmax | 12 hours
AUC(0-inf) | 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Annelize Koch, Principal Investigator — Simbec Orion Ltd
Locations (1):
- Simbec Orion Ltd, Merthyr Tydfil, United Kingdom